CLINICAL TRIAL: NCT02542163
Title: Pilot Evaluation of the NimbleHeart Harness System in Cardiac Rehabilitation (PEN-CR)
Status: Completed | Type: Observational
Sponsor: NimbleHeart Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB #9648
Record Dates: First submitted 2015-08-28; First posted 2015-09-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: To conduct a pilot study to assess the feasibility of the NimbleHeart wireless telemetry vest in cardiac rehabilitation.

Study Design: This is a prospective, single center, non-randomized, pilot trial evaluating the NimbleHeart chest harness system.

DETAILED DESCRIPTION:
20 subjects will be consented to participate at an early cardiac rehabilitation exercise session (typically sessions 1-6). Subjects will wear the NimbleHeart vest concurrently with existing telemetry system during exercise sessions, and thus not replace existing telemetry monitoring. Both staff and subjects will be queried for their (user) experiences during and after each session. Experiences will be documented on surveys after each session. De-identified ECG rhythm strips from the NimbleHeart monitor will be collected to assess quality of tracings. Subjects will be asked to wear the NimbleHeart vest for 2 sessions. Study participation will end after the 2nd session.

ELIGIBILITY:
Inclusion Criteria:

1. Participating in the Cardiac Rehabilitation Program.
2. Capable of giving, and willing to sign, informed consent.

Exclusion Criteria:

1. Patients with either unstable heart disease or unstable heart failure and for whom exercise is contraindicated.
2. Presence of Ventricular Assist Device (VAD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac Rehabilitation phase II population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Degree of difficulty in attaching the harness as compared to attaching the standard telemetry system. | 3 to 4 months
  How "easy" or "difficult" it is to apply the harness system as compared to existing telemetry system.
  Scores range from 1 to 5 scale where 1 = More difficult and 5 = Much easier
Reported occurrences of subject discomfort | 3 to 4 months
  Percentage of subjects with reported harness discomfort and a description of each occurrence of discomfort
Quality of ECG tracings during exercise | 3 to 4 months
  Degree of ECG quality to determine heart rate and detect arrhythmia during subject exercise Scores range from 1 to 3 scale where 1 = Poor and 3 = Good

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States